CLINICAL TRIAL: NCT01856686
Title: Neurocognitive and Neurobiological Improvement in ADHD Children by Modification of Dietary Protein
Acronym: BrainProtein
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Spanish Foundation for Neurometrics Development (Other)
Collaborators: PronoKal Foundation (Other); Child Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Brain Proteins
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: ADD; ADHD
Keywords: ADD; ADHD; Proteins; Dietary; Nutrition; QEEG; ERP; ICA
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BP22042013 (Experimental): This group of patients receive 2.000 kilocalories diet(60 g. carbohydrates, 144 gr of fat and 107 gr of proteins), including 2 protein shakes.
  Interventions: Drug: BP22042013
- Low carbohydrate Diet (Experimental): the second group of patients receive diet of 2.000 Kilo calories without rapidly absorbed carbohydrates and without proteins supplements
  Interventions: Dietary Supplement: Low carbohydrate diet

INTERVENTIONS:
Drug: BP22042013 — This group of patients receive 2.000 kilo-calories diet (60 g. carbohydrates, 144 gr of fat and 107 gr of proteins), including 2 protein shakes.
  Other Names: Brain Proteins Supplements
  Arms: BP22042013
Dietary Supplement: Low carbohydrate diet — the second group of patients receive diet of 2.000 Kilo-calories without rapidly absorbed carbohydrates and without proteins supplements
  Other Names: 2000 Kilo-calories without Fast Absorbing Carbohydrate
  Arms: Low carbohydrate Diet

SUMMARY:
Multicenter, Prospective, randomized, comparative and controlled study about the beneficial effects in behavior and brain connectivity of different dietary patterns in 100 children with ADHD between 7 and 12 years, followed up for 3 months of nutritional therapy.

DETAILED DESCRIPTION:
The investigators collect electroencephalogram (EEG), event related potentials (ERP) data, and behavior parameters in ADD/ADHD children that not take stimulants or other drugs during study. They would only follow some nutritional recommendations based on increasing the amount of dietary protein and fast carbohydrates decrease. The duration of the study will be 6 months, 3 months for recruitment and 3 months for dietary treatment.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosed 12 months before
* no take medication
* BMI above the 25th percentile
* Wiesel score between 80 and 100 (about 120)
* Patients who agree to participate and whose guardians signed the informed consent form

Exclusion Criteria:

* eating disorders
* psychosis, bipolar disorder or depression
* kidney or liver failure
* diabetes
* diuretic or cortisone treatment
* haematological problems
* suprarenal diseases
* cancer
* Brain injury
* Cardiovascular or arrhythmia problems

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moises Aguilar-Domingo, PhD, Principal Investigator — Spanish Foundation for Neurometrics Development
Locations (1):
- New Remedies, Liverpool, Merseyside, United Kingdom

REFERENCES:
- See also: Brainmech Foundation — http://www.bigdata4brain.co.uk

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Carbohydrate Diet: This group of patients receive diet of 2.000 Kilo-calories without rapidly absorbed carbohydrates and without proteins supplements
Period: Overall Study
Arm/Group | BP22042013 | Low Carbohydrate Diet
Started | 31 | 33
Completed | 26 | 22
Not Completed | 5 | 11
Not completed — Lost to Follow-up | 5 | 11

BASELINE CHARACTERISTICS:
Population: All patients without Electroencephalogram recordings at 3 months were excluded from statistical analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | BP22042013 | Low Carbohydrate Diet | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.08 (1.9) | 9.41 (1.87) | 9.23 (1.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 16 | 14 | 30
Reaction time [Mean (Standard Deviation); unit: milliseconds] — Reaction time during visual continuous performance task from 19 channels EEG recordings
  milliseconds | 520.46 (93.27) | 506.59 (65.74) | 514.10 (81.28)
Omission errors [Mean (Standard Deviation); unit: errors] — omission errors during visual continuous performance task from 19 channels EEG recordings (test duration 22 minutes)
  errors | 19.31 (20.69) | 18.00 (15.39) | 18.71 (18.28)
Comission errors [Mean (Standard Deviation); unit: errors] — Comission errors during visual continuous performance task from 19 channels EEG recordings (test duration 22 minutes)
  errors | 4.58 (6.30) | 2.82 (2.79) | 3.77 (5.04)
Occipital alpha waves-frequency [Mean (Standard Deviation); unit: Hz] — Frequency Occipital alpha waves during visual continuous performance task
  Hz | 9.62 (1.02) | 9.48 (0.99) | 9.55 (1.00)
Occipital alpha waves-amplitude [Mean (Standard Deviation); unit: microvolts] — Amplitude of occipital alpha waves during visual continuous performance task
  microvolts | 15.75 (10.45) | 20.56 (17.02) | 17.95 (13.90)
Parietal alpha waves-frequency [Mean (Standard Deviation); unit: Hertz] — Frequency of Parietal alpha waves during visual continuous performance task
  Hertz | 8.72 (1.04) | 9.12 (0.94) | 8.91 (1.00)
Mu wave frequency [Mean (Standard Deviation); unit: Hertz] — Frequency mu waves during visual continuous performance task
  Hertz | 9.07 (1.22) | 9.09 (1.06) | 9.08 (1.14)
Mu waves-amplitude [Mean (Standard Deviation); unit: microvolts] — Amplitude of mu waves during visual continuous performance task
  microvolts | 7.38 (6.77) | 7.87 (8.09) | 7.60 (7.33)
Frontal midline theta activity- frequency [Mean (Standard Deviation); unit: Hertz] | 4.69 (1.13) | 4.88 (1.40) | 4.78 (1.25)
Frontal midline theta activity- amplitude [Mean (Standard Deviation); unit: microvolts] | 8.08 (5.87) | 11.66 (8.17) | 9.72 (7.17)
Monastra ratio [Mean (Standard Deviation); unit: ratio] — Theta wave/ Beta wave ratio
  ratio | 22.15 (8.75) | 25.14 (9.72) | 23.52 (9.23)
weight [Mean (Standard Deviation); unit: Kilograms] | 30.09 (7.66) | 38.15 (11.36) | 33.78 (10.26)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 16.16 (2.87) | 18.77 (3.66) | 17.36 (3.48)
Hyperactivity score (clinical scale) [Mean (Standard Deviation); unit: units on a scale] — Hyperactivity score from clinical questionnaire. Range: minimum value: 0 and maximum value: 8. Higher values represent a worse outcome.
  units on a scale | 3.62 (2.59) | 3.82 (2.67) | 3.71 (2.60)
Impulsivity score (clinical scale) [Mean (Standard Deviation); unit: units on a scale] — Impulsivity score from clinical questionnaire. Range: minimum value: 0 and maximum value: 8. Higher values represent a worse outcome.
  units on a scale | 4.58 (2.42) | 4.82 (2.74) | 4.69 (2.54)
Inattention score (clinical score) [Mean (Standard Deviation); unit: units on a scale] — Inattention score from clinical questionnaire. Range: minimum value: 0 and maximum value: 9. Higher values represent a worse outcome.
  units on a scale | 7.69 (1.52) | 7.91 (1.60) | 7.79 (1.54)
Behavior (clinical scale) [Mean (Standard Deviation); unit: units on a scale] — Behavior assessed by total score of clinical questionnaire (sum of Hyperactivity, Impulsivity and Inattention scores). Range: minimum value: 0 and maximum value: 25. Higher values represent a worse outcome.
  units on a scale | 15.88 (4.95) | 16.55 (5.76) | 16.19 (5.29)

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time at 3 Months
Description: Reaction time during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
milliseconds | 506.58 (108.72) | 510.59 (99.05)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.56593, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.44929, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.81844, Paired t-test

2. Primary Outcome: Omission Errors at 3 Months
Description: Omission errors during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach. (Test duration: 22 minutes)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
errors | 17.15 (19.54) | 14.95 (13.43)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.71152, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.27795, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.47616, Paired t-test

3. Primary Outcome: Comission Errors at 3 Months
Description: comission errors during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach.(Test duration: 22 minutes)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
errors | 2.19 (3.38) | 2.82 (4.05)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.10036, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group changes; Test type: Superiority or Other; p = 0.00820, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 1.00000, Paired t-test

4. Secondary Outcome: Occipital Alpha Waves-frequency at 3 Months
Description: occipital alpha waves-frequency during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
Hz | 9.71 (1.13) | 9.60 (1.24)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.92193, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.50704, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.42314, Paired t-test

5. Primary Outcome: Occipital Alpha Brainwaves Amplitudes at 3 Months
Description: occipital alpha waves amplitudes during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
microvolts | 12.25 (9.89) | 11.99 (11.24)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.08946, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.27795, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.01090, Paired t-test

6. Secondary Outcome: Parietal Alpha Waves-frequency at 3 Months
Description: Parietal alpha waves-frequency during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
Hz | 8.96 (1.09) | 9.21 (1.07)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.73209, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.07965, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.61613, Paired t-test

7. Other Pre Specified Outcome: Weight at 3 Months
Description: Weight after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
kilograms | 31.59 (7.28) | 38.67 (11.18)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.33027, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.00013, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.28019, Paired t-test

8. Secondary Outcome: Mu Wave Frequency at 3 Months
Description: Mu wave frequency during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
Hz | 9.06 (1.13) | 9.07 (1.17)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.94449, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.94574, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.85428, Paired t-test

9. Secondary Outcome: Frontal Midline Theta Activity- Frequency at 3 Months
Description: Frontal midline theta activity- frequency during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
Hz | 4.70 (1.38) | 4.76 (1.30)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.83929, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.97213, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.58323, Paired t-test

10. Primary Outcome: Mu Waves-amplitude at 3 Months
Description: Mu waves-amplitude during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
microvolts | 6.32 (6.38) | 6.05 (5.59)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.05158, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.94574, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.09331, Paired t-test

11. Secondary Outcome: Monastra Ratio at 3 Months
Description: Monastra ratio during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
ratio | 16.88 (9.84) | 22.36 (11.27)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.17383, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.00092, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.15544, Paired t-test

12. Primary Outcome: Frontal Midline Theta Activity- Amplitude at 3 Months
Description: Frontal midline theta activity- amplitude during visual continuous performance task from 19 channels EEG recordings, after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
microvolts | 6.81 (3.62) | 9.13 (7.30)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.39707, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.27945, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.19739, Paired t-test

13. Secondary Outcome: Behavior
Description: Behavior assessed by total score of clinical questionnaire (sum of Hyperactivity, Impulsivity and Inattention scores), after 3 months of nutritional approach.
  Range: minimum value: 0 and maximum value: 25. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
units on a scale | 13.08 (5.11) | 12.45 (5.87)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.50964, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.00710, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.00595, Paired t-test

14. Other Pre Specified Outcome: Body Mass Index at 3 Months
Description: Body mass index after 3 months of dietary approach.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
kg/m2 | 16.50 (2.54) | 18.55 (3.43)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.48336, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.08739, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.37046, Paired t-test

15. Other Pre Specified Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of Participants with Adverse Events as a Measure of Safety and Tolerability of Brain Proteins Supplements
Time Frame: Up to 8 months
Measure: Number; unit: participants
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
participants | 0 | 0

16. Secondary Outcome: Hyperactivity Score
Description: Hyperactivity assessed by clinical questionnaire after 3 months of nutritional approach. Range: minimum value: 0 and maximum value: 8. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
units on a scale | 3.04 (2.39) | 2.68 (2.25)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.45013, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.17374, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.07548, Paired t-test

17. Secondary Outcome: Impulsivity Score
Description: Impulsivity assessed by clinical questionnaire after 3 months of nutritional approach. Range: minimum value: 0 and maximum value: 8. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
units on a scale | 3.96 (2.16) | 3.55 (2.22)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.23226, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.08812, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.00776, Pairedt-test

18. Secondary Outcome: Inattention Score
Description: Inattention assessed by clinical questionnaire after 3 months of nutritional approach. Range: minimum value: 0 and maximum value: 9. Higher values represent a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BP22042013 | Low Carbohydrate Diet
Number analyzed (Participants) | 26 | 22
units on a scale | 6.08 (2.50) | 6.23 (2.43)
Statistical Analysis 1: Comparison: BP22042013 vs Low Carbohydrate Diet; Between-Group Comparison; Test type: Superiority or Other; p = 0.90843, ANCOVA
Statistical Analysis 2: Comparison: BP22042013; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.00413, Paired t-test
Statistical Analysis 3: Comparison: Low Carbohydrate Diet; Within-group comparisons between the baseline and 3 month data; Test type: Superiority or Other; p = 0.00775, Paired t-test

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | BP22042013 | Low Carbohydrate Diet
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 0/26 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes